CLINICAL TRIAL: NCT03063515
Title: Using Acetylcholinesterase Inhibitors to Promote Insulin Secretion in Human Beings
Brief Title: AchE Inhibitor and Insulin
Acronym: AchE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Maria del Pilar Solano, Assistant Professor of Medicine, University of Miami
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20161065
Record Dates: First submitted 2017-02-21; First posted 2017-02-24 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Insulin secretion
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pyridostigmine Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- IVGTT without pyridostigmine (No Intervention): An intravenous glucose tolerance test (IVGTT) will be performed without any medication for baseline comparison.
- IVGTT with pyridostigmine (Active Comparator): An IVGTT will be performed 2 hours after taking one single dose of pyridostigmine 60 mg
  Interventions: Drug: Pyridostigmine

INTERVENTIONS:
Drug: Pyridostigmine — single oral dose of 60 mg pyridostigmine tablet
  Other Names: Mestinon
  Arms: IVGTT with pyridostigmine

SUMMARY:
The investigator will examine the effect of a single dose of pyridostigmine, AchE inhibitor on insulin secretion in healthy subjects. Each subject will undergo an intravenous glucose tolerance test (IVGTT) where IV glucose will be administered and the glucose excursion and insulin secretion response will be evaluated by measuring insulin and glucose at different time points. The test will be carried out twice, once without and once with the administration of a single dose of Pyridostigmine on two separate days. The investigator hypothesizes that inhibiting AChE will potentiate insulin secretion.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older

Exclusion Criteria:

* BMI >30 Kg/m2
* fasting glucose >100
* Glycohemoglobin (Hemoglobin A1C) 5.7% or more
* History of asthma
* Use of medications that may interfere with glucose metabolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
First phase insulin response to IV glucose infusion | -10, -4, 1, 2, 3, 4, 5, 6, 8, and 10 minutes
  Insulin positive incremental area under the curve and the sum of plasma insulin values at 1 minute and 3 minutes after IV glucose infusion

SECONDARY OUTCOMES:
Glucose excursion after IV glucose infusion | -10, -4, 1, 2, 3, 4, 5, 6, 8, and 10 minutes
  Glucose positive incremental area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Pilar Solano, MD, Principal Investigator — University of Miami
Locations (1):
- Diabetes Research Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No